CLINICAL TRIAL: NCT04282954
Title: A Randomized, Double-blind, Active-controlled, Multi-center Phase II Clinical Trial to Evaluate the Safety and Efficacy of JP-1366 in Patients With Erosive Gastroesophageal Reflux Disease
Brief Title: Clinical Trial to Evaluate the Safety and Efficacy of JP-1366 in Patients With Erosive Gastroesophageal Reflux Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Onconic Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JP-1366-201
Record Dates: First submitted 2020-02-21; First posted 2020-02-25 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-07

CONDITIONS: GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): JP-1366 A mg
  Interventions: Drug: JP-1366; Drug: JP-1366 placebo; Drug: Esomeprazole placebo
- Group 2 (Experimental): JP-1366 B mg
  Interventions: Drug: JP-1366; Drug: JP-1366 placebo; Drug: Esomeprazole placebo
- Group 3 (Experimental): JP-1366 C mg
  Interventions: Drug: JP-1366; Drug: JP-1366 placebo; Drug: Esomeprazole placebo
- Goup 4 (Active Comparator): Esomeprazole 40 mg
  Interventions: Drug: JP-1366 placebo; Drug: Esomeprazole 40mg

INTERVENTIONS:
Drug: JP-1366 — JP-1366, QD
  Arms: Group 1; Group 2; Group 3
Drug: JP-1366 placebo — JP-1366 placebo, QD
Drug: Esomeprazole 40mg — Esomeprazole 40mg, QD
  Arms: Goup 4
Drug: Esomeprazole placebo — Esomeprazole placebo, QD
  Arms: Group 1; Group 2; Group 3

SUMMARY:
Clinical trial to evaluate the safety and efficacy of JP-1366 in patients with erosive gastroesophageal reflux disease

ELIGIBILITY:
Inclusion Criteria:

* Adults between 19 and 75 years old based on the date of written agreement
* Those who have been diagnosed with erosive gastroesophageal reflux disease(EGRD) of LA Grade A-D on the upper gastrointestinal endoscopy
* Those who experienced symptoms of heartburn or acid reflux within the last 7 days

Exclusion Criteria:

* Those who have undergone gastric acid suppression or gastric, esophageal surgery
* Those who with clinically significant liver, kidney, nervous system, respiratory, endocrine, hematologic, cardiovascular, urinary system disease
* Clinically significant abnormal laboratory values during screening

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-12-11 (Actual)

PRIMARY OUTCOMES:
Accumulated mucosal defect cure rate*(%) at Week 8 following study drug administration (%) | 8 weeks
  * Erosion recovered to normal mucous membrane on upper gastrointestinal endoscopy

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital and 19 hospitals, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No